CLINICAL TRIAL: NCT06401863
Title: Implementation of DDInteract A Shared-decision Making Tool for Anticoagulant Drug-Drug INTERACTions (DDinteract)
Brief Title: Shared Decision for Drug Interactions in Oral Anticoagulation
Acronym: DDInteract
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Daniel Malone, Professor, University of Utah
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB_00167936; R18HS029300 (AHRQ)
Record Dates: First submitted 2024-04-25; First posted 2024-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Anticoagulants; Drug Interactions
Keywords: Oral anticoagulants; Drug interactions; Gastrointestinal hemorrhage; Shared Decision Making
MeSH Terms: conditions — Gastrointestinal Hemorrhage

STUDY DESIGN:
Intervention Model Description: Rolling implementation at the clinic level with control clinics not exposed to the tool.
Masking Description: No masking due to the nature of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to DDInteract tool in anticoagulated patients (Experimental): This population will consist in outpatient clinics who treat oral anticoagulated patients where DDInteract has been implemented. This intervention is referred to as DDInteract tool exposure in anticoagulated patients. DDInteract may be accessed by clinicians to evaluate risk of harm from drug-drug interactions for patients on anticoagulants.
  Interventions: Other: Shared Decision Making Tool
- Standard of Care (No Intervention): This population will consist in outpatient clinics who treat oral anticoagulated patients where DDInteract has not yet been implemented.

INTERVENTIONS:
Other: Shared Decision Making Tool — EHR-integrated SDM for Patients on Oral Anticoagulants and other medications that might increase the risk of hemorrhage
  Other Names: Shared Decision Making Tool to reduce harm from Drug Interactions
  Arms: Exposure to DDInteract tool in anticoagulated patients

SUMMARY:
The purpose of this project is to implement and evaluate a shared-decision making (SDM) tool called DDInteract that was developed to support decision making for drug-drugs interactions while on oral anticoagulants. DDInteract will be implemented in clinics at the University of Utah, University of Colorado and University of Vanderbilt. DDInteract will be launched from within the electronic health record (EHR) retrieving patient-specific risk factors, will calculate the risk of harm, and will allow providers and patients to dynamically explore "what if" scenarios to optimize treatment and minimize risk. DDInteract will enable shared-decision making using individually-tailored information on the potential benefits and harms of drug interactions in anticoagulated patients.

DETAILED DESCRIPTION:
The purpose of this project are: 1) Examine contextual factors and define relevant implementation strategies to facilitate integration of DDInteract within 3 university-based healthcare systems; 2) Evaluate DDInteract in production/real-world situations to identify barriers and facilitators to adoption and use of DDInteract and to develop solutions to overcome those barriers; 3) Conduct a cluster randomized, multi-system trial to evaluate the effectiveness of DDInteract to mitigate exposure to drug interactions involving oral anticoagulants This project will implement a SDM tool designed to inform clinicians and patients about the risk of harm from drug interactions in patients receiving oral anticoagulants. An initial version of the DDInteract will be EHR-integrated and will be accessed directly in the EHR and auto-populate relevant patient-specific data including other medications that might interact with oral anticoagulants.

This study will use a multi-center randomized cluster design using clinics from the above-mentioned institutions. Each organization will implement DDInteract in their electronic health record system and the study will evaluate the degree to which the tool is utilized within each organization. The implementation period will last 18 months. This project is supported by a R18 award from Agency for Healthcare Research and Quality (AHRQ).

ELIGIBILITY:
Inclusion Criteria:

* Be at least 21 years of age or older
* Receive more than one prescription of an oral anticoagulant (i.e. warfarin, apixaban, edoxaban, dabigatran, rivaroxaban)

Exclusion Criteria:

* Individuals not able to speak English or Spanish

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3691 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Differences of Differences in Estimated Risk of Gastrointestinal Bleeding by DDInteract algorithm | Through study completion, an average of 18 months for the implementation period and 12 months for the baseline period clinics
  We will compare population Gastrointestinal Bleeding risk across the randomized clinics before and after implementation of DDInteract

OTHER OUTCOMES:
Gastrointestinal Bleeding Episodes | Through study completion, an average of 18 months, 6 months per sites (UoU, UC and VU) before and after implementation
  Number of GI hemorrhage episodes by time period in the participation sites before and after DDInteract implementation

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Malone, PhD, Principal Investigator — College of Pharmacy. University of Utah
Locations (3):
- United States (3):
  - University of Colorado. School of Medicine, Denver, Colorado
  - Vanderbilt University, Nashville, Tennessee
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Gomez Lumbreras A, Reese TJ, Del Fiol G, Tan MS, Butler JM, Hurwitz JT, Brown M, Kawamoto K, Thiess H, Wright M, Malone DC. Shared Decision-Making for Drug-Drug Interactions: Formative Evaluation of an Anticoagulant Drug Interaction. JMIR Form Res. 2022 Oct 19;6(10):e40018. doi: 10.2196/40018. PMID 36260377
- [Background] Reese TJ, Del Fiol G, Morgan K, Hurwitz JT, Kawamoto K, Gomez-Lumbreras A, Brown ML, Thiess H, Vazquez SR, Nelson SD, Boyce R, Malone D. A Shared Decision-making Tool for Drug Interactions Between Warfarin and Nonsteroidal Anti-inflammatory Drugs: Design and Usability Study. JMIR Hum Factors. 2021 Oct 26;8(4):e28618. doi: 10.2196/28618. PMID 34698649